CLINICAL TRIAL: NCT06319287
Title: A Phase 2a Multi-Center, Prospective, Randomized Controlled Study to Evaluate the Safety and Efficacy of Topically Applied PEP-TISSEEL in Subjects With Diabetic Foot Ulcers (DFU)
Brief Title: Phase 2a Multi-Center Prospective, Randomized Trial to Evaluate the Safety & Efficacy of Topical PEP-TISSEEL for Diabetic Foot Ulcers (DFU)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rion Inc. (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-00125
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Diabetic Wound; Diabetic Foot; Foot Ulcer; Exosome; Extracellular Vesicle
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Intervention Model Description: Multi-center, Open Label, Randomized Controlled Clinical Trial Evaluating the Effect of PEP/TISSEEL in the Treatment of Diabetic Foot Ulcers
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PEP-TISSEEL+SOC (Active Comparator): Treatment for the PEP-TISSEEL+SOC arm is:
  * PEP-TISSEEL
  * Mepitel dressing followed by Tegaderm® (Mepilex can be used if subjects are allergic to Tegaderm)
  * 3M Cavilon® (may be used on the borders prior to placing the Tegaderm or Mepilex)
  * Padded 3-layer secondary outer layer dressing (Profore (Smith and Nephew (Memphis, TN)); and
  * Offloaded with an offloading Controlled Ankle Movement (CAM) Boot (Foot Defender (Miami, FL) or Total Contact Cast (TCC)) Use of an alternate offloading device (e.g., Charcot Restraint Orthotic Walker (CROW) boot, custom shoe, etc.) may be approved on a case-by-case basis
  Interventions: Biological: PEP (Purified Exosome Product) / TISSEEL
- Standard of Care (Sham Comparator): * Fibracol
  * Mepitel dressing followed by Tegaderm (Mepilex can be used if subjects are allergic to Tegaderm)
  * 3M Cavilon (may be used on the borders prior to placing the Tegaderm or Mepilex )
  * Padded 3-layer secondary outer layer dressing (Profore (Smith and Nephew (Memphis, TN)) or equivalent); and
  * Offloaded with an offloading CAM Boot (Foot Defender (Miami, FL) or TCC)
  * Use of an alternate offloading device (e.g., Charcot Restraint Orthotic Walker (CROW) boot, custom shoe, etc.) may be approved on a case-by-case basis
  Interventions: Biological: PEP (Purified Exosome Product) / TISSEEL

INTERVENTIONS:
Biological: PEP (Purified Exosome Product) / TISSEEL — PEP Drug Product is a lyophilized powder contained within a 10R glass vial. PEP Drug Product is a lyophilized powder derived from apheresed platelets in plasma. The powder cake weighs approximately 75 mg per vial. This protocol will evaluate 2 vials of PEP Drug Product delivered in 10 mL TISSEEL fibrin sealant (15mg/mL PEP-TISSEEL) for 12 weeks.
  TISSEEL is a fibrin sealant indicated as an adjunct to standard surgical techniques (such as suture and ligature) to prevent leakage from colonic anastomoses following the reversal of temporary colostomies
  Other Names: Extracellular Vesicles

SUMMARY:
This is a Phase 2a Multi-Center, Prospective, Randomized, Controlled Study aimed to evaluate the Safety and Efficacy of Topically Applied PEP-TISSEEL in Subjects with Diabetic Foot Ulcers (DFU)

DETAILED DESCRIPTION:
The objective of this multi-center, prospective, randomized controlled study is to evaluate the safety and efficacy of PEP-TISSEEL+ Standard of Care (SOC) compared to SOC only treatment in up to 60 subjects (30 subjects PEP-TISSEEL + SOC and 30 subjects SOC only), specifically for the treatment of their non-healing DFU.

Treatment for the PEP-TISSEEL+SOC arm is:

* PEP-TISSEEL
* Mepitel dressing followed by Tegaderm® (Mepilex can be used if subjects are allergic to Tegaderm)
* 3M Cavilon® (may be used on the borders prior to placing the Tegaderm or Mepilex)
* Padded 3-layer secondary outer layer dressing (Profore (Smith and Nephew (Memphis, TN)); and
* Offloaded with an offloading Controlled Ankle Movement (CAM) Boot (Foot Defender (Miami, FL) or Total Contact Cast (TCC))

  * Use of an alternate offloading device (e.g., Charcot Restraint Orthotic Walker (CROW) boot, custom shoe, etc.) may be approved on a case-by-case basis

Treatment for the Standard of Care (SOC) only arm is:

* Fibracol
* Mepitel dressing followed by Tegaderm (Mepilex can be used if subjects are allergic to Tegaderm
* 3M Cavilon (may be used on the borders prior to placing the Tegaderm or Mepilex)
* Padded 3-layer secondary outer layer dressing (Profore (Smith and Nephew (Memphis, TN)) or equivalent); and
* Offloaded with an offloading CAM Boot (Foot Defender (Miami, FL) or TCC)

  * Use of an alternate offloading device (e.g., Charcot Restraint Orthotic Walker (CROW) boot, custom shoe, etc.) may be approved on a case-by-case basis

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Properly obtained written informed consent
3. Documented history of Type I or Type II Diabetes Mellitus, requiring oral and/or insulin replacement therapy
4. The index ulcer is classified as Wagner grade 1 ulcer and remains Wagner 1 Grade between Screening and Randomization/Baseline visit (Visit 1 through Visit 3)
5. These ulcers are superficial, full-thickness ulcers limited to the dermis, not extending to the subcutaneous tissue
6. Area of index ulcer must be between 1 cm2 to 15 cm2 post debridement at screening and baseline
7. The index ulcer must be located anatomically on the foot with ≥ 50% of the wound area below the medial or lateral malleolus
8. Presence of a persistent nonhealing DFU for at least 4 weeks from Randomization and not more than 1 year that has failed to respond to SOC at any point during this timeframe
9. Adequate vascular perfusion as evidenced by one of the following:

   1. Dorsal transcutaneous oxygen measurement (TCOM/TcPO2) measurement of

      ≥ 40 mmHg within 90 days of Screening (Visit 1 or 2)
   2. Ankle Branchial Index (ABI) between 0.7 and 1.3 within 90 days of Screening (Visit 1 or 2) using the extremity on which the index ulcer is located
   3. Arterial Doppler ultrasound evaluating for biphasic or triphasic dorsalis pedis and/or posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable within 90 days of Screening (Visit 1 or 2)
10. The index ulcer has been offloaded with protocol defined offloading device during Screening (Run-In) period through Randomization/Baseline visit.
11. Must meet one of the following criteria:

    a. Female subjects of Non-Child-Bearing Potential defined as: i. Postmenopausal for at least 1 year (Subject verbal confirmation acceptable), or surgically sterilized (i.e., hysterectomy or bilateral oophorectomy more than 3 months prior to Screening (Visit 1 or 2)), or ii. Bilateral tubal ligation more than 6 months prior to Screening (Visit 1 or 2), or iii. Must have a negative serum β-hCG pregnancy test at Visit 1 and not be breastfeeding prior to being administered with the study drug b. Male subjects of Non-Childbearing Potential are defined as those vasectomized subjects whose vasectomy was performed 6 months prior to Screening (Visit 1 or 2) or those diagnosed as sterile by a physician c. Females and Males of Childbearing Potential who practice an acceptable method of contraception defined as the use of any form of hormonal contraceptive, a barrier method with spermicide, condoms, intrauterine device, or abstinence from sexual intercourse starting at least 60 days prior to Screening and continuing at least 30 days following the last treatment.

    Female will undergo a negative serum β-hCG pregnancy test at Visit 1 and an additional urine test at Baseline/Randomization (Visit 3 or Day 0) and must not be breastfeeding prior to being administered with the study drug
12. Ability to comply with the study protocol as per investigator discretion

Exclusion Criteria:

1. Actively undergoing chemotherapy treatment (localized radiation treatment is allowed if it is not on the DFU wound site and in remission based on scans, bloodwork or some other kind of test, such as a breast biopsy or a bone marrow biopsy)
2. Ulceration with exposed tendon, capsule, or bone
3. Suspicion of bone or joint infection by clinical or other criteria as per STONEES criteria below:

   a. STONEES criteria for infection: i. size increase, ii. temperature elevation, iii. os (probe to bone) iv. new areas of breakdown v. exudative vi. erythema/edema vii. smell
4. Unable or unwilling to utilize the protocol defined offloading device
5. Subjects who have undergone endovascular or open revascularization of the index limb within the last 30 days from Screening.
6. Index ulcer has decreased in area by ≥ 30% between Screening (Visit 1) and Baseline visits
7. Any subject that is currently on/or requires oral, systemic or topical antibiotics, or is anticipated to require their use during the course of the study
8. Any subject that has vascular compromise requiring surgical intervention or has undergone vascular reconstruction or angioplasty less than 1 month prior to randomization. Any planned surgical procedures during the study participation
9. Serum Creatinine level > 3.0 mg/dL
10. Hemoglobin A1c (HbA1c) >12%
11. Aspartate Aminotransferase (AST, GOT) and/or Alanine Aminotransferase (ALT, GPT) >3x the upper limit of normal
12. Acute active Charcot foot
13. The location of the index ulcer is within 2 cm of any other ulcer
14. Any subject that would be unable to safely monitor the infection status of the index ulcer at home and return for scheduled visits
15. History of immunosuppression or taking immunosuppressive agents including systemic corticosteroids, except stable daily doses of 5 mg/day or less for chronic conditions for up to 5 days
16. Any subject with a life expectancy ≤ 6 months
17. Pregnancy, including a positive pregnancy test at Baseline, or lactation/breastfeeding at anytime
18. Use of investigational drugs or biologics within 28 days prior to screening (Visit 1 or 2)
19. History of a concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol
20. Known or suspected active abuse of alcohol, or non-prescription drugs
21. Participation in another interventional clinical study or study in the past 30 days of Screening (Visit 1 or 2) or concurrent participation in another interventional clinical study
22. Subjects who have untreated Hep C
23. Subjects who are HIV positive
24. Subjects on anticoagulation that are not maintained within the International Normalized Ratio (INR) of > 3.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 12 weeks
  Complete wound closure (wound healing) by 12 weeks (efficacy; landmark analysis)
Safety | 6 months
  Count dose limiting toxicity events (incidence of treatment-emergent adverse event)

SECONDARY OUTCOMES:
Percent Area Reduction of Wound at 12 Weeks | 12 weeks
  Percentage area reduction (PAR) at 12 weeks.

OTHER OUTCOMES:
Visual Analogue Scale (VAS) for Pain over 12 weeks | 12 weeks
  VAS pain (mean difference between baseline and 12 weeks) from 0 (No Pain) to 10 (Worst Possible Pain)
Semmes-Weinstein Score | 12 weeks
  Semmes-Weinstein score (mean difference between baseline and 12 weeks)
Wound-Q Scale | 12 weeks
  Wound-Q (domains: wound characteristics and health-related quality of life; mean difference between baseline and 12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Professional Education & Research Institute (PERI), Blue Ash, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rion company website — https://riontx.com/about/
- See also: PERI company website — https://www.periedu.com/